CLINICAL TRIAL: NCT05134389
Title: Survey on Gastrointestinal and Nutritional Parameters Among One Anastomosis Gastric Bypass Patients From Different Countries
Brief Title: Survey on GI and Nutritional Parameters Among OAGB Patients From Different Countries
Status: Completed | Type: Observational
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Shiri Sherf Dagan, Dietitian and Epidemiologist, Principal Investigator, Assuta Medical Center
Other Study IDs: ASMC-0104-19
Record Dates: First submitted 2021-11-13; First posted 2021-11-26 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Obesity
Keywords: bariatric surgery; gastric bypass; weight outcomes; functional gastrointestinal disorders; nutrition
MeSH Terms: conditions — Obesity; Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Israel: OAGB patients from Israel
  Interventions: Procedure: One Anastomosis Gastric Bypass
- Spain: OAGB patients from Spain
  Interventions: Procedure: One Anastomosis Gastric Bypass
- Portugal: OAGB patients from Portugal
  Interventions: Procedure: One Anastomosis Gastric Bypass

INTERVENTIONS:
Procedure: One Anastomosis Gastric Bypass — Exposure to One Anastomosis Gastric Bypass

SUMMARY:
One Anastomosis Gastric Bypass (OAGB) surgery is a type of bariatric surgery (BS) which is gaining popularity worldwide and is considered to be a simple, safe and effective bariatric procedure in terms of weight loss and comorbidities resolution. However, only limited data exists on the nutritional and gastrointestinal (GI) consequences of this procedure.

This study aimed to gain information on GI and nutritional parameters from a large sample of OAGB patients living in 3 different countries.

Post-OAGB patients across Israel (n=277), Spain (n=105) and Portugal (n=111) were recruited to the study based on the time elapsed since surgery [1-6 months (1-6M), 6-12 months (6-12M) and 1-5 years (1-5Y) post-surgery]. Participants were asked to complete an anonymous survey delivered by SurveyMonkey®️ software which included data on demographics, comorbidities, anthropometrics, GI outcomes and satisfaction with the procedure.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years old
* patients who underwent primary OAGB in the last 5 years

Exclusion Criteria:

* patients who had undergone other bariatric surgery
* current pregnancy
* lacked capacity to consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or above who underwent primary OAGB in the last 5 years from Israel, Spain and Portugal
Sampling Method: Non-Probability Sample
Enrollment: 493 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Self-reported anthropometric outcomes | Only once in accordance to the time group (1-6 months, 6-12 months and 1-5 years post-surgery).
  Measured by weight changes

SECONDARY OUTCOMES:
A. Self-reported lifestyle outcomes | Only once in accordance to the time group (1-6 months, 6-12 months and 1-5 years post-surgery).
  Measured by satisfaction and quality of life scales (scale of 0-100)
B. Self-reported lifestyle outcomes | Only once in accordance to the time group (1-6 months, 6-12 months and 1-5 years post-surgery).
  Measured by attendance to follow-up regime (no. of meetings)
C.Self-reported lifestyle outcomes | Only once in accordance to the time group (1-6 months, 6-12 months and 1-5 years post-surgery).
  Measured by adherence to the bariatric surgery health recommendations [physical activity (min/week), alcohol drinking (doses/day), smoking (current/past/never) and supplementation usage (non/monthly/weekly/daily)]
A. Self-reported nutritional outcomes | Only once in accordance to the time group (1-6 months, 6-12 months and 1-5 years post-surgery).
  Measured by adherence to the bariatric surgery eating recommendations questionnaire (0=no, 1=partial, 2=yes)
B. Self-reported nutritional outcomes | Only once in accordance to the time group (1-6 months, 6-12 months and 1-5 years post-surgery).
  Measured by taste change, smell change and food aversion questionnaire (yes/no/open text for additional information)
C. Self-reported nutritional outcomes | Only once in accordance to the time group (1-6 months, 6-12 months and 1-5 years post-surgery).
  Measured by self-reported questionnaire for quick assessment of food tolerance after bariatric surgery (scored between 1-27, while higher scores represents better tolerance)
A. Self-reported GI outcomes | Only once in accordance to the time group (1-6 months, 6-12 months and 1-5 years post-surgery).
  Measured by no. defecations per day and defecations texture
B. Self-reported GI outcomes | Only once in accordance to the time group (1-6 months, 6-12 months and 1-5 years post-surgery).
  Measured by severity of dyspepsia symptoms scale (4-point graded scale -0 represents absence of symptoms and 3 represents severe symptoms which interfere to perform normal activities)
C. Self-reported GI outcomes | Only once in accordance to the time group (1-6 months, 6-12 months and 1-5 years post-surgery).
  Measured by Gastrointestinal Symptom Rating Scale (GSRS) (scored 15-105, while higher scores represents more severe symptoms)

CONTACTS AND LOCATIONS:
Locations (1):
- Assuta Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided